CLINICAL TRIAL: NCT03245138
Title: Endoscopic Third Ventriculostomy Versus Ventriculo-peritoneal Shunting in Idiopathic Normal Pressure Hydrocephalus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Principal Investigator, Sascha Marx, Principal Investigator, University Medicine Greifswald
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ETV versus VPS in iNPH
Record Dates: First submitted 2017-07-31; First posted 2017-08-10 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Normal Pressure Hydrocephalus
Keywords: endoscopic third ventriculostomy; ventricular peritoneal shunt; communicating hydrocephalus
MeSH Terms: conditions — Hydrocephalus, Normal Pressure; Hydrocephalus | interventions — Ventriculostomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- endoscopic third ventriculostomy (Experimental): endoscopic third ventriculostomy for the treatment of iNPH
  Interventions: Procedure: Endoscopic Third Ventriculostomy
- ventricular peritoneal shunt (Active Comparator): Insertion of a ventriculo-peritoneal Shunt for the treatment of iNPH
  Interventions: Procedure: Ventriculo-Peritoneal Shunting

INTERVENTIONS:
Procedure: Endoscopic Third Ventriculostomy — patients receive an endoscopic third ventriculotomy as surgical procedure
  Arms: endoscopic third ventriculostomy
Procedure: Ventriculo-Peritoneal Shunting — patients receive an ventriculo-peritoneal shunt as surgical procedure
  Arms: ventricular peritoneal shunt

SUMMARY:
An endoscopic third ventriculostomy is considered to be successful in idiopathic normal pressure hydrocephalus (iNPH) in some literature reports, but there is a lack of high quality data. The aim of the present study is to compare the treatment options of iNPH (Endoscopic third ventriculostomy versus ventriculo-peritoneal shunt) in a randomized, controlled, multicenter study.

DETAILED DESCRIPTION:
The traditional treatment for communicating hydrocephalus is a ventriculo-peritoneal shunt insertion and the endoscopic third ventriculostomy (ETV) is reserved for patients with obstructive hydrocephalus. However, in the last decade several reports highlighted an success of an ETV in communicating hydrocephalus as well. Thus, the aim of the present study is to compare ventriculo-peritoneal shunting against ETV in patients with an idiopathic normal pressure hydrocephalus, an subset of communicating hydrocephalus, in a randomized, controlled multicenter study.

ELIGIBILITY:
Inclusion Criteria:

* Age over 50 years
* gait disturbances typical for iNPH
* symptoms Duration less than 36months
* exclusion of obstructive hydrocephalus
* positive spinal TAP-test

Exclusion Criteria:

* no informed consent
* malignant disease
* other diseases of the CNS (Parkinson, dementia)
* secondary communicating hydrocephalus

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Kiefer Index | 1 year
  Improvment of at least 2 points
Recovery Index | 1 year
  Improvment of at least 2 points

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - University Medicine Göttingen, Göttingen
  - University Medicine Greifswald, Greifswald
  - Klinikum Neubrandenburg, Neubrandenburg

IPD SHARING:
Plan to Share IPD: Undecided